CLINICAL TRIAL: NCT02226653
Title: A Bioequivalence and Food Effect Study of Evacetrapib Evaluating a Single Tablet Compared to Two Tablets in Healthy Japanese Subjects
Brief Title: A Study of Evacetrapib in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14627; I1V-JE-EIAY (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (reference) (Experimental): Single oral dose of 1 tablet of evacetrapib on Day 1 of up to three of five periods
  Interventions: Drug: Evacetrapib
- Evacetrapib (test) (Experimental): Single oral dose of 2 tablets of evacetrapib on Day 1 of up to three of five periods
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595

SUMMARY:
The purpose of this study is to determine if two different dosing strategies for evacetrapib will have essentially the same effect on the body. The study will also explore the effect of a low fat meal on how the body absorbs evacetrapib. This study will last at least 15 weeks, not including screening. Screening is required within 28 days prior to the date of first dosing.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese, as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.0 to 29.9 kg/m^2
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal supine blood pressure as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Are women who are pregnant or lactating
* Have used or intend to use over-the-counter, prescription medications, or herbal medicine 14 days prior to enrollment and during the study
* Have donated blood of more than 400 mL in the last 12 weeks (males) or in the last 16 weeks (females), or any blood donation (including apheresis) within the last 4 weeks
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to abide by alcohol restrictions
* Are participants who currently smoke more than 10 cigarettes per day or are unwilling to abide by smoking restrictions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Periods 1 to 4 participants are in the fasting state and Period 5 participants were fed a low fat meal. There were two fixed sequences for Test (T) and Reference (R) doses with each participant receiving 5 doses. There was a washout period of at least 21 days between doses.
Groups:
- Reference/Test/Reference/Test/Test: Reference (R) dose is a single oral dose of one - 130 mg tablet of evacetrapib on Day 1 of Period 1 and Day 1 of Period 3. Test (T) dose is a single oral dose of Test two - 65 mg tablets of evacetrapib on Day 1 of Period 2, Day 1 of Period 4 and Day 1 of Period 5. There was a washout period of at least 21 days between doses.
- Test/Reference/Test/Reference/Reference: Test (T) dose is a single oral dose of two - 65 milligram (mg) tablets of evacetrapib on Day 1 of Period 1 and Day 1 of Period 3. Reference (R) is a single oral dose of Reference (R) one - 130 mg tablet of evacetrapib on Day 1 of Period 2, Day 1 of Period 4 and Day 1 of Period 5. There was a washout period of at least 21 days between doses.
Period: Treatment Period 1 Fasted State
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 24 | 24
Received at Least 1 Dose of Study Drug | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Washout Period 1 (at Least 21 Days)
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Treatment Period 2 Fasted State
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 24 | 24
Received at Least 1 Dose of Study Drug | 24 | 24
Completed | 23 | 24
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout Period 2 (at Least 21 Days)
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Treatment Period 3 Fasted State
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Received at Least 1 Dose of Study Drug | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Washout Period 3 (at Least 21 Days)
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Treatment Period 4 Fasted State
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Received at Least 1 Dose of Study Drug | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Washout Period 4 (at Least 21 Days)
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Treatment Period 5 Fed State
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 24
Received at Least 1 Dose of Study Drug | 23 | 24
Completed | 23 | 23
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout Period 5 (at Least 21 Days)
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Reference/Test/Reference/Test/Test: Reference(R) dose is a single oral dose of Reference 1 one- 130 mg tablet of evacetrapib on Day 1 of Period 1 and Day 1 of Period 3. Then, Test (T) dose is a single oral dose of Test 2 two- 65 mg tablets of evacetrapib on Day 1 of Period 2, Day 1 of Period 4 and Day 1 of Period 5. There was a washout period of at least 21 days between doses.
- Test/Reference/Test/Reference/Reference: Test (T) dose is a single oral dose of Test 2 two- 65 mg tablets of evacetrapib on Day 1 of Period 1 and Day 1 of Period 3. Then, Reference (R) dose is a single oral dose of Reference 1 one- 130 mg tablet of evacetrapib on Day 1 of Period 2, Day 1 of Period 4 and Day 1 of Period 5. There was a washout period of at least 21 days between doses.
- Total: Total of all reporting groups
Arm/Group | Reference/Test/Reference/Test/Test | Test/Reference/Test/Reference/Reference | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.9) | 34.7 (11.3) | 33.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 24 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve From Zero to Infinity (AUC[0-∞]) of Evacetrapib (Fasted)
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 Hours Post-dose in Periods 1,2,3, and 4
Population: All randomized participants who completed and had evaluable AUC(0-∞) bioequivalence fasted state data for Periods 1,2,3 and 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram·hour/milliliter (ng·h/mL)
Groups:
- Reference (Fasted): Reference dose is a single oral dose of Reference one- 130mg tablets of evacetrapib in fasted state in Period 1, 2, 3 and 4.
- Test (Fasted): Test dose is a single oral dose of Test two- 65mg tablets of evacetrapib in fasted state in Periods 1, 2, 3 and 4.
Arm/Group | Reference (Fasted) | Test (Fasted)
Number analyzed (Participants) | 45 | 45
nanogram·hour/milliliter (ng·h/mL) | 14600 (40) | 14600 (36)

2. Primary Outcome: PK: Maximum Concentration (Cmax) of Evacetrapib (Fasted)
Time Frame: as for outcome 1
Population: All randomized participants who completed and had evaluable Cmax bioequivalence fasted state data for Periods 1,2,3 and 4.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Reference (Fasted) | Test (Fasted)
Number analyzed (Participants) | 45 | 45
nanogram/milliliter (ng/ml) | 1130 (53) | 1100 (40)

3. Secondary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of Evacetrapib (Fasted and Fed)
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 Hours Post-dose in Periods 2,4, and 5
Population: All randomized participants who completed and had evaluable Tmax Fasted and Fed State data for Periods 2, 4, and 5.
Measure: Median (Full Range); unit: hour (h)
Groups:
- Reference (Fasted): Reference dose is a single oral dose of Reference one- 130mg tablets of evacetrapib in fasted state in Periods 2 and 4.
- Reference (Fed): Reference dose is a single oral dose of Reference one- 130mg tablets of evacetrapib in fed state in Period 5.
- Test (Fasted): Test dose is a single oral dose of Test two- 65mg tablets of evacetrapib in fasted state in Periods 2 and 4.
- Test (Fed): Test dose is a single oral dose of Test two- 65mg tablets of evacetrapib in fed state in Period 5.
Arm/Group | Reference (Fasted) | Reference (Fed) | Test (Fasted) | Test (Fed)
Number analyzed (Participants) | 23 | 23 | 22 | 22
hour (h) | 3.75 [1.75 to 5.00] | 2.50 [1.50 to 5.50] | 3.50 [2.25 to 5.00] | 2.75 [2.00 to 6.00]

4. Secondary Outcome: PK: AUC(0-∞)of Evacetrapib (Fasted and Fed)
Time Frame: as for outcome 3
Population: All randomized participants who completed and had evaluable AUC(0-∞) Fasted and Fed State data for Periods 2,4, and 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Groups:
- Reference (Fed): Reference dose is a single oral dose of Reference one- 130mg tablets of evacetrapib in fed state in Periods 5.
Arm/Group | Reference (Fasted) | Reference (Fed) | Test (Fasted) | Test (Fed)
Number analyzed (Participants) | 23 | 23 | 22 | 22
ng·h/mL | 14800 (39) | 18900 (24) | 14600 (39) | 18600 (26)

5. Secondary Outcome: PK: Cmax of Evacetrapib (Fasted and Fed)
Time Frame: as for outcome 3
Population: All randomized participants who completed and had evaluable Cmax Fasted and Fed State data for Periods 2,4, and 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Reference (Fasted) | Reference (Fed) | Test (Fasted) | Test (Fed)
Number analyzed (Participants) | 23 | 23 | 22 | 22
ng/ml | 1100 (57) | 1450 (21) | 1090 (44) | 1480 (27)

ADVERSE EVENTS:
Description: The safety population includes all 48 participants who enrolled in the study.
Groups:
- 130 mg Tablet Evacetrapib (Fasted): Reference dose is a single oral dose of Reference one- 130 mg tablets of evacetrapib in fasted state in Periods 1, 2, 3, and 4.
- 2 x 65 mg Tablets Evacetrapib (Fasted): Test dose is a single oral dose of Test two- 65mg tablets of evacetrapib in fasted state in Periods 1, 2, 3, and 4.
- 130 mg Tablet Evacetrapib (Fed): Reference dose is a single oral dose of Reference one- 130 mg tablets of in fed state in Period 5.
- 2 x 65 mg Tablets Evacetrapib (Fed): Test dose is a single oral dose of Test two- 65mg tablets of evacetrapib in fed state in Period 5.
Arm/Group | 130 mg Tablet Evacetrapib (Fasted) | 2 x 65 mg Tablets Evacetrapib (Fasted) | 130 mg Tablet Evacetrapib (Fed) | 2 x 65 mg Tablets Evacetrapib (Fed)
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/48 | 2/48 | 0/23 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 130 mg Tablet Evacetrapib (Fasted) (N=48) | 2 x 65 mg Tablets Evacetrapib (Fasted) (N=48) | 130 mg Tablet Evacetrapib (Fed) (N=23) | 2 x 65 mg Tablets Evacetrapib (Fed) (N=23)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days